CLINICAL TRIAL: NCT07000799
Title: Coping@School: A Study of School Absenteeism and Student Well-being in Elementary Schools
Brief Title: A Study of School Absenteeism and Student Well-being in Elementary Schools
Acronym: Coping@school
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Kristin Kicki Martinsen, Professor in Psychology, PhD, University of Oslo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 853141; 853141 (Other: Regional Committees for Medical and Health Research Ethics)
Record Dates: First submitted 2025-04-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: School Absenteeism; Anxiety and Depression
Keywords: school absenteism; anxiety; depression; Prevention; Early intervention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm with new groups entering the intervention every semester (Experimental): The design is a single arm pre-post design where the children will receive the EMOTION intervention over 8 weeks and attendance teams will be implemented in their school. The EMOTION Intervention is based on cognitive-behavioral therapy, which has been shown to be effective in both the treatment and prevention of anxiety and depression in children. The EMOTION intervention has been developed as a school-based program and consists of an intensive course lasting eight weeks, using a hybrid model with eight face-to-face group meetings at school and eight hours of digital sessions completed by the child at home. Additionally, it is desirable for parents to support their children; hence, guardians will be offered the opportunity to attend an informational meeting. They will also receive a brochure detailing how they can support and assist their child. A group leader manual and a workbook for the children have been developed (Martinsen et al., 2017).
  In the children's groups, participants
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — The EMOTION Intervention is based on cognitive-behavioral therapy, which has been shown to be effective in both the treatment and prevention of anxiety and depression in children. The EMOTION intervention has been developed as a school-based program and consists of an intensive course lasting eight weeks, using a hybrid model with eight face-to-face group meetings at school and eight hours of digital sessions completed by the child at home. Additionally, it is desirable for parents to support their children; hence, guardians will be offered the opportunity to attend an informational meeting. They will also receive a brochure detailing how they can support and assist their child. A group leader manual and a workbook for the children have been developed (Martinsen et al., 2017).

SUMMARY:
This study will be conducted at elementary schools in Oslo and aims to explore multiple aspects of school absenteeism and student well-being. It has two main objectives: 1) a preventive focus specifically related to school attendance and functioning, and 2) a user perspective that includes measuring user satisfaction with the interventions used in the study. The aim is to investigate whether the EMOTION intervention can be utilized to enhance school attendance and functioning for children experiencing emerging difficulties in attending school, who also tend to be more sad and anxious than their peers. Additionally, the study seeks to compare changes in anxiety and sadness with previous studies involving the EMOTION intervention through benchmarking. The perceptions of parents regarding the causes of their children's difficulties will also be examined. Evaluating user satisfaction with the EMOTION intervention in relation to emerging school absenteeism and the implementation of attendance teams in the schools is another objective. This will contribute to increased knowledge about interventions targeting children with emerging difficulties in school attendance and their experiences with these interventions.

DETAILED DESCRIPTION:
School absenteeism is a growing problem among children and youth, often associated with complex and varied causes. Anxiety and sadness are common challenges for children and can impact their functioning in many areas, including school performance. Early intervention regarding anxiety and sadness in a school context can be crucial for improving students' school experience and coping skills. The EMOTION intervention has been tested in two randomized controlled trials, where the intervention group showed a significant reduction in symptoms of anxiety and sadness compared to the control group. However, the intervention has not been investigated in relation to school attendance in larger studies. Furthermore, since 2017, several primary schools in Oslo have established interdisciplinary attendance teams. Assessing user satisfaction with these teams is essential for improving efforts with children struggling with school attendance. Thus, the Coping@School study aims to undertake a comprehensive mapping and evaluation of interventions that may contribute new knowledge in addressing emerging issues related to school attendance.

GENERAL BACKGROUND School Absenteeism In a Norwegian study of students in grades 6 to 10 across seven municipalities, 3.6% reported that their absenteeism was related to school refusal. This indicates that at least one student in every class shows signs of school refusal or is at risk of developing it. Schools and PPT report a rise in school refusal, according to, and other studies suggest that problems related to school absenteeism begin early in a student's educational journey (Hancock et al., 2013). Absenteeism can result from the school environment (such as social belonging, motivation, bullying, teaching methods, and teacher support), familial factors (such as parents' mental health and involvement), and individual factors concerning the child (for example, low self-esteem and emotional difficulties such as anxiety or sadness). Patterns of absenteeism are established and escalate over time, contributing to increasing knowledge gaps and symptoms of emotional distress. Belonging to school, friends, and self-confidence in solving challenging situations may thus diminish. It is therefore essential to identify challenges early so that a negative trajectory can be reversed before negative patterns are established and school attendance is difficult.

In a report, it is mentioned that academic challenges and school-related stress are among the factors influencing students' absenteeism. This can diminish opportunities for education and future income. According to Sintef (2012), school absenteeism can also lead to socioeconomic costs if it results in a lack of connection to the labor market in adulthood. The societal economic costs due to school dropout were estimated at approximately five billion Norwegian kroner for each annual cohort in Norway in 2010. A more recent economic analysis from 2021 revealed that social exclusion, defined as high school dropout rates, costs Norway a minimum of 73 billion annually due to lost income, benefits, and premature death. Addressing school absenteeism is therefore critical from a socioeconomic perspective in addition to the consequences it has for individuals.

The new education act has introduced stricter requirements for following up on absenteeism. Among the most important changes is the obligation for municipalities and counties to ensure that students with absenteeism from education are followed up. This obligation applies to all absenteeism, starting from the first day a student is absent from instruction. Effective systems and routines for registering various types of absenteeism, identifying absenteeism patterns, following up on absent students, and cooperating with families must be in place. The follow-up of absenteeism must be tailored to the cause, duration, and frequency. Interventions may be necessary for children who are sad or anxious, as this can also contribute to difficulties with school attendance. This must be considered in light of the education act, particularly Chapter 12 concerning school environment and Chapter 10 addressing adapted education and individual adjustments.

The national professional guidelines for school health services for youth emphasize that school health services should collaborate with schools to plan and implement initiatives that promote well-being and health. School-based interventions targeting risk factors for absenteeism are therefore vital. School health services should be involved early in following up on students with concerning absenteeism and can provide interventions aimed at triggering difficulties such as anxiety and sadness. Anxiety and Sadness Anxiety disorders rank among the most common mental health issues among children and youth, with estimates suggesting that between 5.6% and 18.1% of children may develop an anxiety disorder before they turn 18.. Depression likewise represents a prevalent condition among children and youth, with estimates of between 1-2% of children and between 3-8% of adolescents likely to experience this condition. Studies also suggest that between 9-12% of children exhibit symptoms of anxiety and depression that interfere with daily functioning, even if they do not meet the criteria for diagnosis. Both problems represent a significant public health concern. The challenges associated with anxiety and depression negatively impact children across many areas of life, potentially complicating their relationships with peers and family members. A close relationship exists between anxiety and school absenteeism. In studies examining school refusal, it is common for between 50% and 60% of participants to meet criteria for an anxiety disorder, with an even greater number experiencing sub-threshold symptoms. Sadness and depression are similarly prevalent among those struggling with school attendance; in a population study, 14% of school refusers also had a diagnosis of depression. Sub-threshold symptoms such as sleep difficulties and fatigue/loss of energy were also prevalent.

Research indicates that anxious and sad children and adolescents are less likely to receive help than children with externalizing disorders. Implementing interventions within the school setting offers an opportunity to identify and reach children who might otherwise receive little assistance for their challenges. Should this approach increase school attendance and reduce potential dropout, several crucial societal missions would be fulfilled.

The EMOTION intervention is an evidence-based intervention aimed at children exhibiting elevated levels of anxiety and/or depression symptoms. The program has been evaluated in two randomized controlled trials, demonstrating significant reductions in symptoms for participating children.

Relationship Between School Attendance/Functioning and Anxiety/Sadness Given the correlation between participation and functioning at school and anxiety/sadness, it is essential to investigate if an intervention like EMOTION could also contribute to the reduction of problems associated with school attendance, improve school functioning, while simultaneously maintaining reductions in symptoms of anxiety and sadness as demonstrated in previous studies. To date, only a pilot study (N = 4) has been conducted exploring whether anxious and sad children also show improved school attendance following participation in a mastery group. Results from this study are summarized in a thesis at the Department of Psychology, University of Oslo, indicating a reduction in reported school refusal behaviors after participating in the intervention, as reported by both the children themselves and their parents. This suggests increased school attendance following participation in the mastery group. However, testing interventions for children with emerging school absenteeism is still novel and has been seldom explored in previous research. Existing studies primarily focus on children and youth with established difficulties with school absenteeism. Gaining insights into the efficacy of this intervention concerning school attendance, school functioning, and symptoms of emotional distress is therefore vital. This study will also incorporate user satisfaction to further evaluate the interventions. Assessing user satisfaction in relation to both such interventions and attendance teams in schools is a new approach that aims to provide a more comprehensive understanding of the measures targeting children with emerging difficulties in school attendance. This way, the study will contribute valuable knowledge in addressing the needs of this group of children.

MAIN OBJECTIVES OF THE STUDY Objectives The primary objective of the study is twofold, encompassing a preventive perspective and a user perspective. Within the preventive perspective, the goal is to conduct coping groups aimed at children who are beginning to experience difficulties related to school attendance and who exhibit higher levels of anxiety and sadness than their peers. The study seeks to evaluate changes in school attendance and functioning, as well as in anxiety and/or sadness. Moreover, it aims to explore the potential reasons behind these challenges from the parents' perspective. The user perspective will be assessed by mapping user satisfaction related to both the coping groups (reported by children, parents, and group leaders) and the attendance teams at schools (reported by teachers, professionals in PPT/school health services, and school leadership). Throughout the study, a comprehensive understanding of interventions aimed at addressing emerging difficulties in school attendance will be achieved.

Research Questions:

1 a) Will children participating in a coping groups demonstrate increased school attendance and improved school functioning immediately following the intervention (T2) and after six months (T3) compared to baseline (T1)?

1. b) Will children participating in a coping group report comparable changes in symptoms of anxiety and/or sadness as reported by parents, children, and teachers, immediately following the intervention (T2) and after six months (T3) compared to previous studies of the intervention (benchmarking)?
2. a) How do parents, children, and group leaders evaluate their satisfaction with participation in the coping group aimed at increasing school attendance?

2 b) To what extent are participants in the attendance team (contact teachers, school leaders, school health services, counselors in special education services) satisfied with the function and use of the attendance team? 3) What are parents' perceptions of the causes of their children's difficulties with school attendance, and what support and assistance do they seek from the school and other agencies? DESIGN AND METHODS Design This study will employ a one-group pretest-posttest design to examine changes in school attendance and functioning, as well as changes in symptoms of anxiety and sadness before and after the intervention is implemented. User satisfaction with the EMOTION intervention aimed at enhancing school attendance, as well as with the attendance team, will also be investigated.

Children aged 9 to 13 years (grades 4 to 7) (N = 112) who are struggling with school attendance and functioning and exhibit slightly higher levels of anxiety and sadness than their peers (see also Section 3.3 below) will be invited to participate in the coping groups at elementary schools in Oslo. All schools will implement an attendance team to monitor school attendance and absences. The children will be assessed for participation prior to the coping group, immediately after the intervention, and six months later (see detailed assessment procedures below).

Procedure for Identification and Selection of Participants The identification and selection of children will be based on experiences from the evaluations conducted of the EMOTION intervention through two randomized controlled studies (Martinsen et al., 2019; Neumer et al., 2021; Patras et al., 2016) and the most recently conducted pilot study related to school absenteeism. All studies have been approved by the Regional Committee for Medical and Health Research Ethics for South-Eastern Norway (REK Sør-Øst; approvals 2013/1909, 2019/1198, and REK ID 639838, February 2024). It will be communicated to teachers, parents, and children that participation is voluntary. Participants sought for recruitment to the pilot project are children aged 9 to 13 years (grades 4 to 7) who display early difficulties related to school participation/functioning and exhibit slightly higher levels of anxiety and sadness than their peers. Thus, they may be at risk of developing problems related to school attendance, as well as escalating levels of anxiety and sadness.

Information and Informed Consent:

1. Recruitment begins with a meeting involving the school administration, social worker, and grade-level teachers for the relevant classes (grades 4-7). During this meeting, professionals from the Psychological - Educational-Services (PPT) in Oslo will provide information about the study and emphasize the importance of ensuring that parents and students do not feel pressured to participate; participation is entirely voluntary.
2. Parents will receive information about the study at a parent meeting, and subsequently, all parents in the grade will receive information about the study, both written and electronically. Interested parents can then attend a digital parent meeting for more specific information regarding the study and the initiative. Students will also be presented with information about the project in class, along with age-appropriate information regarding the study. Both the presentation and written materials will emphasize that participation is voluntary. Information for children and guardians will be distributed via the school's standard communication channels (digitally).
3. Both parents must provide written informed consent for children who wish to participate to be assessed in the next phase.
4. Students in the relevant grade level who wish to participate and have consent from both guardians will be evaluated in the next phase. Children at this age do not have the capacity to consent, but it is nonetheless important that their voices are heard. The information letter to guardians about the initiative will therefore encourage parents to discuss potential participation with their children and ensure that children are heard if they do not wish to participate. This is in line with recommendations from the Ethical Committee in previous studies of the initiative, including the pilot study. It will be made clear to parents at this stage, and at any later point, that participation is voluntary and that they have the option to withdraw their child from participation in the support group and the study at any time.
5. Assessment: Children who express interest in participating and have consent from both guardians will respond to questions related to early school absenteeism (SCREEN and self-developed questions) (see measurement instruments below). They will also respond to questions regarding anxiety and sadness (RCADS). The survey will be administered electronically at school with a teacher present. The chosen questionnaire, RCADS (see measurement instruments below), in which the child self-assesses their symptoms, is increasingly used in both clinical and non-clinical samples in relation to preventive measures and demonstrates good psychometric properties among Norwegian children. Parents will fill out a similar questionnaire to that of their children in the parent version and will additionally answer questions regarding possible causes of school absenteeism (SRAS), as well as self-developed questions related to school attendance and functioning. The same will apply to contact teachers who have selected students for the support group, who will respond to similar questions related to school participation and functioning, as well as record attendance/absenteeism.

Follow-up for Children Not Offered the Support Group: Information will be provided both at the parent meeting and when children are introduced to the initiative in class that the group will consist of maximum 7 children in the coping group each semester, and that children in need who may not get an invitation will have priority in the following semesters should their issues persist. If there are more eligible children than available in the group, those offered a place will be determined through a random selection (randomization procedure). If parents and the child want such help, those not offered a group placement will be followed up by the school's attendance team, and if other support is needed beyond the school health service, or relevant support agencies connected to the school will be contacted.

Procedure for Identifying Special Needs: Children who, for various reasons, would not benefit from a group intervention-such as those with low cognitive abilities or children with developmental disorders-will be evaluated individually for participation. The project will be conducted in collaboration with the school health service and the Educational-Psychological Services (PPT), and robust follow-up procedures will be established if the assessment reveals children with concerning levels of symptoms, specific plans for suicide, and/or other circumstances indicating an urgent need for assistance. If PPT identifies children in the group who raise concerns, the project team's group leaders will promptly contact the guardians and, if applicable, the school administration and local PPT representatives to discuss further actions and possible evaluations concerning the child.

Recruitment Plan and Scope: Data collection will take place over four semesters (spring and fall 2025, spring and fall 2026, spring 2027). The plan is to include up to seven children receiving the coping group interventions from 1st to 2nd grades each semester (Spring 2025: 6th and 7th grades; Fall 2025: 6th grade; Spring 2026: 5th grade; Fall 2026: 4th grade). Children will be assessed before the intervention and immediately after its completion. In addition, they will complete the same questionnaires six months after the intervention has ended..

The school's overall absenteeism data for grades 1-7 will be collected between November 2024 and January 2025 to establish a baseline for absenteeism at the school, as well as in spring/fall 2025, spring/fall 2026, and spring 2027 to evaluate whether the combination of the attendance team and the Empowering Children groups leads to reduced absenteeism.

The initiative will be implemented in elementary schools in Oslo that have voluntarily expressed their interest in participation.

Resources: The Oslo PPT has allocated resources to provide information in schools as well as to lead the groups (two active professionals and three trained professionals available for support as needed). The Health Agency in Oslo collaborates with the Oslo PPT to deliver information at the selected schools. Additionally, the school health nurse will be involved. A strong partnership has been established with the relevant schools, which will also appoint a contact person for the study. A research assistant/data handler will assist in data collection using Nettskjema, and they, along with psychology students from the professional program at the Psychological Institute, will conduct qualitative interviews with two to three parents at each participating school. The project lead from PSI/UIO will oversee the coordination of the project.

The EMOTION intervention The EMOTION Intervention is based on cognitive-behavioral therapy, which has been shown to be effective in both the treatment and prevention of anxiety and depression in children. The EMOTION intervention has been developed as a school-based program and consists of an intensive course lasting eight weeks, using a hybrid model with eight face-to-face group meetings at school and eight hours of digital sessions completed by the child at home. Additionally, it is desirable for parents to support their children; hence, guardians will be offered the opportunity to attend an informational meeting. They will also receive a brochure detailing how they can support and assist their child. A group leader manual and a workbook for the children have been developed (Martinsen et al., 2017). Several studies have been conducted of the EMOTION intervention , including the ECHO study (2020 - 2023) (Neumer et al., 2021), the TIM study (2013 - 2017) (Patras et al., 2016), a pilot study (2012 - 2013) (Martinsen et al., 2016), and a pilot study of "Mestrende barn" and school attendance in 2024 (REK ID 639838).

Data Management Since the project leader at PSI receives royalties from the sale of materials, the recruitment of schools and participants, as well as data management, will be conducted by individuals within or associated with the project who have no conflicts of interest. Data will be collected and stored through the Services for Sensitive Data (TSD) at the University of Oslo, which meets the stringent legal requirements for the processing and storage of sensitive research data in a secure project area. Consequently, the data will be stored on a password-protected server with restricted access. All data will be stored in accordance with the University of Oslo's guidelines and ethical standards.

Group Leaders, Training, and Supervision The intervention will be carried out by qualified health personnel working in the school health service and in PPT Oslo. The group leaders have received training in the EMOTION program through a two-day course as well as a two-hour course covering the digital module. Supervision will be provided when coping groups are running.

Collaboration The project has been established in collaboration with Oslo PPT, led by senior advisor Lise Sæhle (project leader 1), the Health Authority of Oslo Municipality, with special consultant Gudrun Abel Engh (project leader 2), and Professor Kristin Martinsen at the Department of Psychology UiO (project leader 3), forming the project management team. Furthermore, collaboration has been established with leaders of the school health service in the municipalities involved as well as with the principals of the four participating schools. All participating schools have signed collaboration agreements for the study.

Professionals from RKBU Midt-Norge/NTNU, led by Associate Professor Jo Magne Ingul, and the University of Stavanger, National Center for School Environment and Behavioral Research, represented by Professor Trude Havik, play an advisory role in the project and are also members of a steering committee alongside the data protection officer at the Department of Psychology, UiO, Torgrim Langleite.

The primary working group consists of professionals from PPT Oslo, the Health Authority in Oslo, and UiO. Responsibility for project management is distributed among PPT Oslo, the Health Authority, and the University of Oslo to ensure that the project is implemented and communicated in an objective and credible manner. The project group will also include a research assistant/data manager who will work 20% of their time to develop the online survey for data collection and conduct qualitative interviews alongside psychology students from the Department of Psychology, UiO. Additionally, an independent statistician will be associated with the project group to conduct independent analyses of the collected data to ensure objective and credible data representation.

EXPECTED BENEFITS OF THE STUDY It is anticipated that the project, through systematic interdisciplinary collaboration and development, will provide municipal services with knowledge about the use of evidence-based methods to increase school attendance among sad and anxious children. This could improve the overall quality of services while providing necessary assistance to children and parents specifically. Through the project, children who otherwise would not receive help will be reached, and provisions will be made for making the initiative available to more children with similar needs in the future. The project will also contribute knowledge to the field regarding early intervention for children facing difficulties related to school attendance.

TIMELINE Timeline: The project will be conducted January 1, 2025, to June 30, 2027. ETHICS AND DATA PROTECTION Analysis of responses will only be conducted on anonymized data and will be carried out by an independent statistician with no conflicts of interest in the project. The project is conducted in accordance with the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* Children wherer the child or parents report difficulties related to school participation/functioning
* and who exhibit elevated symptom levels for self-reported anxiety and/or sadness RCADS - 47

Exclusion Criteria:

* Children who are deemed not to benefit from a group intervention includeing children with low cognitive capacity or with developmental disorders.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primar outcomes for absenteeism | From screening for enrollment (T1), at the end of treatment after approximately 10 weeks (T2) and 6 moths after the intervention finished (T3)
  Primary outcome measures Children:
  School attendance: Screen for Early Development of School Absenteeism: SCREEN. Scores from 1 - 5 , not at all to very, higher score indicates higher absentism.
  Primary outcome measures Parents:
  Screen for Early Development of School Absenteeism: SCRE

CONTACTS AND LOCATIONS:
Overall Officials: Kristin D. Martinsen, PhD, Principal Investigator — UiO
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
At this time, we do not have definitive plans to share Individual Participant Data (IPD) with other researchers due to several considerations. Firstly, we are committed to maintaining participant confidentiality and adhering to data protection regulations, which may restrict the international sharing of data. Additionally, the study still in its early stages, and we are assessing the feasibility and ethical implications of data sharing as the project progresses.
  We recognize the importance of data sharing for advancing research and may explore opportunities for future collaboration that align with ethical guidelines and regulatory requirements. Should circumstances change, we will develop a transparent sharing plan that ensures compliance with applicable laws and safeguards participant confidentiality.

REFERENCES:
- [Background] Martinsen KD, Rasmussen LMP, Wentzel-Larsen T, Holen S, Sund AM, Lovaas MES, Patras J, Kendall PC, Waaktaar T, Neumer SP. Prevention of anxiety and depression in school children: Effectiveness of the transdiagnostic EMOTION program. J Consult Clin Psychol. 2019 Feb;87(2):212-219. doi: 10.1037/ccp0000360. Epub 2018 Dec 13. PMID 30550301